CLINICAL TRIAL: NCT06333483
Title: A Single-Arm, Open-Label, Phase I Study to Determine the Safety, Tolerability and Preliminary Efficacy of Obecabtagene Autoleucel in Patients With Severe, Refractory Systemic Lupus Erythematosus
Brief Title: Obe-cel in Adolescent [Applicable in UK Only] and Adult Severe, Refractory Systemic Lupus Erythematosus
Acronym: CARLYSLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO1-SL1; 2023-508236-60-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-06; First posted 2024-03-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: AUTO1; Obecabtagene autoleucel (obe-cel); CD19-positive chimeric antigen receptor T cell; CAR-T
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AUTO1 (Experimental)
  Interventions: Biological: Obecabtagene autoleucel (obe-cel)

INTERVENTIONS:
Biological: Obecabtagene autoleucel (obe-cel) — Following lymphodepletion with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with a single dose of obe-cel

SUMMARY:
This is a Phase 1 study of obecabtagene autoleucel (obe-cel), autologous T cells engineered with a chimeric antigen receptor (CAR) targeting CD19, to establish the tolerability, safety, preliminary efficacy, and pharmacokinetics of obe-cel in patients with severe, refractory SLE.

DETAILED DESCRIPTION:
This is a single-arm, open-label Phase 1 Study to determine the safety, tolerability, and preliminary efficacy of obe-cel in patients with severe, refractory SLE. Up to a maximum of 18 patients will be treated in a maximum of 3 dose levels.

By using the Bayesian Optimal Interval (BOIN) design for overdose control, the Sponsor will review the Safety Review Committee (SRC) and Independent Data Monitoring Committee (IDMC) recommendation and determine if a dose level is suitable for a subsequent study.

ELIGIBILITY:
Inclusion Criteria:

-Key Inclusion Criteria-

* Women or men ≥ 18 years at screening [Spain only] or patients 12 to 65 years of age (inclusive) at the time of signing the informed consent [UK only]
* Diagnosis of SLE fulfilling the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) Classification Criteria for Systemic Lupus Erythematosus
* Positive for at least one of the following autoantibodies: antinuclear antibodies (ANA) at a titer of ≥ 1:80, or anti-dsDNA (≥ 30 IU/mL) or anti-Smith (> upper limit of normal [ULN]), anti-histone or anti-chromatin (> ULN)
* Severe, refractory SLE

Exclusion Criteria:

-Key Exclusion Criteria-

* Medications

  * Within 2 months of leukapheresis: use of anti-CD20 therapy
  * Prior treatment with anti-CD19 therapy (including bispecifics), adoptive T cell therapy or any prior gene therapy product (e.g., CAR T cell therapy)
  * Immunization with a live or attenuated vaccine within 2 months of leukapheresis
* SLE and Autoimmunity:

  * Recurrent neuropsychiatric lupus or active, severe or unstable neuropsychiatric lupus within 2 years from screening
  * Diagnosis of drug-induced SLE rather than idiopathic SLE
  * Any acute, severe lupus-related flare during screening that needs immediate treatment and/or makes the immunosuppressive washout impossible; thus, making the patient ineligible for CD19 CAR T therapy as judged by the Investigator or Sponsor
  * Significant, likely irreversible organ damage related to SLE (e.g., end-stage renal disease) that in the opinion of the Investigator renders CD19 CAR T cell therapy unlikely to benefit the patient
  * Diagnosis of another non-SLE autoimmune disease (e.g., dermatomyositis, polymyositis, scleroderma, rheumatoid arthritis) or overlap syndrome
* Medical History:

  * History or presence of: (Within 3 months before screening visit)

    * Clinically relevant central nervous system (CNS) pathology such as epilepsy, paresis, aphasia, or stroke
    * Evidence of deep venous thrombosis or pulmonary embolism
  * History or presence of severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, uncontrolled mental illness, or psychosis
  * Clinically significant, uncontrolled heart disease not due to SLE (New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled cardiac arrhythmia, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless the patient has a pacemaker) or a recent (within 12 months of screening) cardiac event
  * Active or uncontrolled fungal, bacterial, viral (including COVID-19), or other infection requiring systemic antimicrobials for management
  * Active or latent hepatitis B or active hepatitis C
  * Human immunodeficiency virus, human T-cell leukemia virus (HTLV)-1, HTLV-2 or syphilis positive test at screening
  * History of malignant neoplasms unless disease free for at least 24 months (basal cell or squamous cell carcinoma in situ, or in situ breast cancer on hormonal therapy allowed)
  * History of heart, lung, kidney, liver transplant or hematopoietic stem cell transplant
  * Pregnancy or lactating
* Laboratory and Organ Function:

  * Left ventricular ejection fraction < 45% (or < institute's lower limit of normal) confirmed by echocardiogram
  * Oxygen saturation (SpO2) < 90% in the absence of oxygen support
  * B cell aplasia

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | Up to 28 days from obe-cel infusion
  Percentage of patients receiving obe-cel who experience dose-limiting toxicities (DLTs)
Adverse events | Up to Month 12
  Adverse event (AE) type, frequency, severity, and relationship with obe-cel and lymphodepletion of AEs

SECONDARY OUTCOMES:
Remission rate according to Definition of Remission in SLE (DORIS) | Up to Month 12
  Remission rate as specified by Definition of Remission in SLE (DORIS)
Response over time according to Definition of Remission in SLE (DORIS) | Up to Month 12
  Response over time as specified by Definition of Remission in SLE (DORIS)
Time to response according to Definition of Remission in SLE (DORIS) | Up to Month 12
  Time to response as specified by Definition of Remission in SLE (DORIS)
Change over time in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | Up to Month 12
  Change compared to baseline in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score. The total score is the sum of all marked SLE-related descriptors. A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Change over time in Physician's global assessment (PGA) | Up to Month 12
  Change compared to baseline in physician's global assessment (PGA) of average SLE disease severity on a visual analog scale (VAS) between 0 and 3 where 0 represents no disease, 1 represents mild disease activity, 2 represents moderate disease activity, and 3 represents a severe disease activity (highest and most severe possible disease activity). At least 10% change improvement or worsening in PGA to be clinically significant compared to baseline
Pharmacokinetics (maximum serum concentration [Cmax]): Detection of CAR-T cells by polymerase chain reaction (PCR) in peripheral blood | Up to Month 12
  Detection of CAR T cells measured by PCR in the peripheral blood after obe-cel infusion
Pharmacokinetics (time to reaching maximum serum concentration [Tmax]): Detection of CAR-T cells by polymerase chain reaction (PCR) in peripheral blood | Up to Month 12
  Detection of CAR T cells measured by PCR in the peripheral blood after obe-cel infusion
Pharmacokinetics (area under the curve [AUC]): Detection of CAR-T cells by polymerase chain reaction (PCR) in peripheral blood | Up to Month 12
  Detection of CAR T cells measured by PCR in the peripheral blood after obe-cel infusion
Pharmacokinetics (last observed quantifiable concentration [Clast]): Detection of CAR-T cells by polymerase chain reaction (PCR) in peripheral blood | Up to Month 12
  Detection of CAR T cells measured by PCR in the peripheral blood after obe-cel infusion
Pharmacokinetics (time to reach last observed quantifiable concentration [Tlast]): Detection of CAR-T cells by polymerase chain reaction (PCR) in peripheral blood | Up to Month 12
  Detection of CAR T cells measured by PCR in the peripheral blood after obe-cel infusion
Pharmacodynamics: B cell aplasia | Up to Month 12
  Depletion of circulating B cells in the peripheral blood

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (2):
  - Hospital Universitari Vall Hebrón, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - Addenbrookes Hospital, Cambridge
  - University College London Hospitals NHS Foundation Trust, London
  - Great Ormond Street Hospital, London
  - Manchester Royal Infirmary, Manchester University NHS Foundation Trust,, Manchester